CLINICAL TRIAL: NCT03170921
Title: Psychophysiological Characterization of Different Capoeira Performances in Experienced Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alfredo Anderson Teixeira de Araujo (Other)
Responsible Party: Sponsor-Investigator, Alfredo Anderson Teixeira de Araujo, Master of Science, Universidade Federal do vale do São Francisco
Organization: Universidade Federal do vale do São Francisco (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: UFSaoFrancisco3_
Record Dates: First submitted 2017-05-20; First posted 2017-05-31 (Actual); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Physical Activity; Affective; Reaction; Physiological Stress
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Angola (Experimental): The rhythm performance had duration of 90 seconds. During recovery period (post- intervention) in the moments 1, 3, 5, 7, and 9 minutes was measured the physiological and the perceptual variables of the study.
  Interventions: Other: Angola
- Benguela (Experimental): The rhythm performance had duration of 90 seconds. During recovery period (post- intervention) in the moments 1, 3, 5, 7, and 9 minutes was measured the physiological and the perceptual variables of the study.
  Interventions: Other: Benguela
- São Bento (Experimental): The rhythm performance had duration of 90 seconds. During recovery period (post- intervention) in the moments 1, 3, 5, 7, and 9 minutes was measured the physiological and the perceptual variables of the study.
  Interventions: Other: São Bento

INTERVENTIONS:
Other: Angola — The rhythm performance (Angola) had duration of 90 seconds. During recovery period (post- intervention) in the moments 1, 3, 5, 7, and 9 minutes was measured the physiological and the perceptual variables of the study.
  Arms: Angola
Other: Benguela — The rhythm performance (Benguela) had duration of 90 seconds. During recovery period (post- intervention) in the moments 1, 3, 5, 7, and 9 minutes was measured the physiological and the perceptual variables of the study.
  Arms: Benguela
Other: São Bento — The rhythm performance (São Bento) had duration of 90 seconds. During recovery period (post- intervention) in the moments 1, 3, 5, 7, and 9 minutes was measured the physiological and the perceptual variables of the study.
  Arms: São Bento

SUMMARY:
The aim of this study was to characterize the psychophysiological demand in different Capoeira performances in male experienced individuals. Eleven men healthy and experienced in Capoeira. Participants were invited to five visits in different days: 1) anamnesis and anthropometric assessment; 2) aerobic performance assessment; 3 to 5) performance of 90s in three Capoeira styles (Angola, Benguela and São Bento). Main Outcome Measure(s): The physiological demand through the heart rate (HR), R-R interval (RRi), blood pressure (BP), blood lactate ([Lac]), and glucose ([Gluc]) and rating perceived effort (RPE), feeling scale (FS) and perceived activation (PA) were assessed after 10min of rest and during recovery (1, 3, 5, 7 and 9min) of each performance. HR and RRi records also occurred during each performance.

DETAILED DESCRIPTION:
The present study was approved by the Research Ethics Committee from the Federal University of Vale do São Francisco - UNIVASF under number 1.687.330. The study had as inclusion criteria: (i) to be male between 18 and 40 years; (ii) a Capoeira practitioner for at least 2 years; and (iii) mastering the technique of the three rhythms of performance investigated (Angola, Benguela and São Bento). As exclusion criteria: (i) to be hypertensive, diabetic or obese; (ii) a smoker; (iii) alcohol addicted and (iv) have some cardiovascular dysfunction or musculoskeletal problem. The participants volunteered and signed a written informed consent in accordance with resolution 466/12 from the National Health Council of Brazil and principles of the Declaration of Helsinki. Finally, the sample was composed of 11 male individuals with experience in the three rhythms of Capoeira performance selected for the study. For the evaluation of aerobic fitness was a Maximal Aerobic Incremental Test (MAIT) in the cyclergometer was performed (Biotec 2100, Cefise). MAIT began with one minute warm-up without load, with 50 watts or power followed by increments of 25 watts of power to each stage of one minute. The participants were instructed to maintain a frequency of 50 rpm's during the entire test, until voluntary exhaustion or not maintaining the pre-established rotation. The last stage of the test was considered valid when the individual remained at least 50% of the stage time duration in exercise. During the MAIT, measures of aerobic power, RPE and HR were obtained. The Capoeira performance experimental sessions were performed based on three distinct rhythms, namely: 1) Angola; 2) Benguela and; 3) São Bento. The choice of these performance rhythms is justified because they are the most practiced in the Capoeira world and the literature has reported possible differences in technical standards of physical requirement between them. The performance rhythms were performed in different days and separated by an interval of 48 hours. All the performance rhythms were accompanied by standardized percussion instruments, with three berimbaus, one with severe intonation (berimbau gunga), another intermediate (medium berimbau) and the last with acute intonation (berimbau viola), an atabaque and two tambourines. The musical instruments were played by experienced individuals and the songs were also sung in a standardized way for each performance. The performances in different rhythms always occurred at the same time of day between 3:00 and 4:00 p.m. A period of rest (pre-intervention) with a duration of 10 minutes occurred prior to completion of each performance rhythm, with volunteers being seated comfortably in an upholstered armchair. At the end of the rest measurements of the physiological and the perceptual variables of the study were performed. Soon after the pre-intervention a standardized warm-up/stretching in light intensity perceived was performed during 5 minutes with the own Capoeira movements. Then pairs of participants were conducted for the intervention with the performing of its respective Capoeira performance rhythms (Angola, Benguela or São Bento). Each rhythm of performance had duration of 90 seconds and participants received voice instructions to start and finish the performance. After each physical performance with the Capoeira rhythm, during recovery period (post- intervention) in the moments 1, 3, 5, 7, and 9 minutes was measured the physiological and the perceptual variables of the study. The pre-intervention, intervention and post-intervention were performed in a room free of noise and temperature between 22-24ºC. During the experimental sessions the participants used a device brand Polar Electro Oy mod. RS800CX duly validated to record the HR and R-R intervals (RRi) of HR variability (HRV). In addition to the analysis pre- and post-intervention, during the intervention it was considered the lowest HR and RRi (MIN), the average HR and RRi (AVE) and the largest HR and RRi (PEAK). The records of the RRi, during the intervention, were exported from the device Polar to the software Polar ProTrainer 5 by infra red and analyzed through the software Kubios HRV version 2.0. In order not to jeopardize the reliability of the indexes obtained, the early ectopic and artifact beats were removed and adjusted, being a criterion the differences greater than 20% in relation to adjacent beats. After editing the RRi, analyzes using linear methods in the time and frequency domain were performed with the objective of estimation of cardiac autonomic modulation. Concerning the time domain, the parameters analyzed were the absolute mean RRi and rMSSD (root mean square differences of successive RRi) as an indicator of the modulation of the parasympathetic nervous system. As to frequency domain the high frequency components (HF: 0.15 to 0.4 Hz) as well as the low frequency (LF: 0.04 to 0.15 Hz) were analyzed to calculate the LF:HF ratio, which characterizes the cardiac sympathovagal balance In the pre- and post-intervention BP measures were conducted by means of an automatic sphygmomanometer brand Microlife, mod. BP3AC1-1PC, equipment validated and with high reproducibility for normotensive individuals. The procedures adopted for BP evaluation were those recommended by the Cardiology Brazilian Society. Besides, in the pre- and post-intervention periods a puncture in the participants' ear lobe was done to collect 25 μl of capillary blood by calibrated capillaries. The blood samples were deposited in Eppendorf microtubules and stored in 50 μl of sodium fluoride to 1% for later analysis of [Lac] and [Gluc]]. To this end, a biochemistry electroenzymatic analyzer (Yellow Springs 2,700 STAT, OH, USA) was properly calibrated and used. During MAIT and at the pre- and post-intervention periods with the experimental sessions the perceptual variables were measured through psychometric scales. Rate of perceived exertion (RPE): The whole-body perceived exertion was assessed using the Borg's RPE [6-20] Scale. Before the MAIT, and experimental sessions with Capoeira, the meaning of RPE was explained to the subjects. A rating of 6 (low anchor, "very, very light") was assigned to the lowest exercise intensity, while a rating of 20 (high anchor, "very, very hard") was assigned to the highest exercise intensity. Basic affective response: The Feeling Scale (FS) was used to assess the affective response and it is an 11-point bipolar scale ranging from +5 to -5, commonly used to measure pleasure/displeasure during exercise. This scale presents the following verbal anchors: -5 = very bad; -3 = bad; -1 = fairly bad; 0 = neutral; +1 fairly good; +3 = good; and +5 = very good. The subjects received standard instructions regarding to the use of the FS in according to Hardy and Rejeski. Perceived activation (PA): The PA scale was used to assess the arousal state of the participants. The PA scale is a 6-point single-item measure, ranging from +1 (low arousal) to +6 (high arousal). This scale assesses how the participant felt activated, stimulated and motivated during different times of the study (pre- and post-intervention). In addition, an integrated analysis interpolating FS and PA responses was performed, aiming to obtain the sense that the affective domain points from different quadrants of the circumplex model (high activation-pleasure; high activation-displeasure; low activation-displeasure; low activation-pleasure). Finally, standard definitions of perceptual responses and separate instructional sets for scales were read to the participants immediately before the MAIT. The low and high perceptual anchors for the RPE, FS and PA scale were established during the MAIT. RPE, FS and PA values were evaluated randomly during the last 10 seconds of each stage of MAIT, during pre-intervention and, different moments of post-intervention. Descriptive statistics with mean and standard deviation was performed. The normality of data distribution was tested by the Shapiro-Wilk test. ANOVA two-way for repeated measures, reporting the "F-ratio", degrees of freedom and the "P" value was used to verify the interaction time*rhythms and the main effect of time within each Capoeira performance. The test of Mauchly was adopted to verify the sphericity of the data, which, in case of violation, the degrees of freedom would be corrected by the epsilon of Greenhouse-Geisser. Partial eta squared (ηp2) was used to determine the effect size. Post hoc of Bonferroni was adopted for identification of pairs of difference. The alpha was set at 5% and the software used was SPSS 22.0 for Windows (SPSS, Inc., Chicago, IL).

ELIGIBILITY:
Inclusion Criteria:

* to be male between 18 and 40 years;
* a Capoeira practitioner for at least 2 years;
* mastering the technique of the three rhythms of performance investigated (Angola, Benguela and São Bento).

Exclusion Criteria:

* to be hypertensive, diabetic or obese;
* to be a smoker;
* alcohol addicted;
* have some cardiovascular dysfunction or musculoskeletal problem.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2016-09-05 (Actual); Primary Completion 2016-09-12 (Actual); Study Completion 2016-09-16 (Actual)

PRIMARY OUTCOMES:
Physiological responses (Heart rate) | 30 minutes
  Heart rate (bpm) responded differently among the three investigated rhythms.
Physiological responses (heart rate variability) | 30 minutes
  Heart rate variability indicator, R-R interval (ms), responded differently among the three investigated rhythms.
Physiological responses (Blood lactate) | 30 minutes
  Blood lactate (mmol/L) responded differently among the three investigated rhythms.
Physiological responses (Blood glucose) | 30 minutes
  Blood glucose (mg/dL) responded differently among the three investigated rhythms.

SECONDARY OUTCOMES:
Psychological responses (Rate of perceived exertion response) | 30 minutes
  Rate of perceived exertion response exhibited differences when analyzed the São Bento performance in comparison to the Angola and Benguela performances in Capoeira.
Psychological responses (Basic affective response) | 30 minutes
  Basic affective response exhibited differences when analyzed the São Bento performance in comparison to the Angola and Benguela performances in Capoeira.
  The Feeling Scale (FS) was used to assess the affective response and it is an 11-point bipolar scale ranging from +5 to -5, commonly used to measure pleasure/displeasure during exercise.7 This scale presents the following verbal anchors: -5 = very bad; -3 = bad; -1 = fairly bad; 0 = neutral; +1 fairly good; +3 = good; and +5 = very good. The subjects received standard instructions regarding to the use of the FS.

IPD SHARING:
Plan to Share IPD: No
No.